CLINICAL TRIAL: NCT03687008
Title: Cognitive Intervention to Improve Working Memory in Adolescents With Single Ventricle Heart Disease
Brief Title: Cognitive Intervention to Improve Working Memory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Nancy Pike, PhD, RN, Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 92418
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Single Ventricle Heart Disease
Keywords: Cognition; Working Memory; Magnetic Resonance Imaging; Cogmed

STUDY DESIGN:
Intervention Model Description: one group, pre- post-intervention design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescents with SVHD (Experimental): All adolescents will receive the intervention Cogmed. This is an in home, computer based, cognitive intervention to improve working memory, supervised by trained coaches, [25 sessions, each 30-45 minutes, 5 days a week / 5 week duration].
  Interventions: Behavioral: Cognitive Computer Based Intervention

INTERVENTIONS:
Behavioral: Cognitive Computer Based Intervention — 25 sessions [each 30-45 minutes, 5 days a week / for 5 weeks], supervised by trained coaches
  Other Names: Cogmed Version 4.0

SUMMARY:
Adolescents with single ventricle heart disease (SVHD) (10 males and 10 females) with mild to moderate cognitive impairment will participate in a total of 25 computer-based working memory training sessions, each 30-40 minutes (5 days a week for 5 weeks) supervised by a trained coach. Primary objective is to evaluate the impact of the Cogmed intervention on working memory scores and the secondary objective to assess brain tissue changes with magnetic resonance imaging (MRI) using diffusion tensor imaging (DTI) techniques, measures of mean diffusivity pre- and post-intervention.

DETAILED DESCRIPTION:
Adolescents with single ventricle heart disease (SVHD) show brain injuries in sites (hippocampus, mammillary bodies, thalamus, and frontal cortices) that are associated with cognitive deficits, in particular working memory. A key component of cognition, and thus, an important influence on academic performance, self-care ability, quality of life, and morbidity and mortality, is working memory. However, it is unclear whether cognition, as well as brain tissue integrity can be improved with cognition intervention. Among available interventions, a possible intervention to improve working memory and brain status in SVHD is Cogmed®, which is an interactive, computer-based intervention, specifically designed for children and young adults, to improve attention and working memory with significant effectiveness in other pediatric conditions associated with brain injury. A unique feature of the Cogmed ® program is the in-home support of trained coaches for the duration of the intervention (5 days/week for 5 weeks), which optimizes adherence and confirms completion of the tasks. The investigators will use a one group pre- post-intervention design, 20 subjects (10 males and 10 females), with inclusion criteria: 14-18 years of age, have undergone surgical palliation, and score 25-10 (mild to moderate cognitive impairment) on the Montreal Cognitive Assessment (MoCA) screener. Using non-invasive brain magnetic resonance imaging (MRI) procedures, diffusion tensor imaging (DTI) based mean diffusivity (MD), an MRI measure of tissue integrity, can identify changes in the hippocampus, mammillary bodies, thalamus, and frontal cortices pre- and post- cognitive intervention. Therefore, the specific aims of this proposal are to: 1) examine the impact of Cogmed® intervention on working memory (working memory index [WMI] score from the WRAML2) in adolescents with SVHD (pre- and post-intervention); 2) assess the effect of Cogmed® on brain structural integrity (DTI-based MD procedures) in sites that control memory (hippocampus, mammillary bodies, thalamus, and frontal cortices) in adolescents with SVHD (pre- and post-intervention); and 3) examine if there is an impact of the Cogmed® intervention on cognition and brain tissue integrity based on sex in SVHD.

In summary, SVHD adolescents have significant cognitive deficits that are linked to brain injury in regions, which control such functions. Intervention to improve cognition and brain injury in SVHD is unclear, but a potential innovative treatment for such symptoms and brain injury is Cogmed®. The information from this pilot study has the potential to revolutionize the clinical treatment specific to cognitive deficits in SVHD and other types of congenital heart defects. In addition, the clinical implications are considerable as improved working memory skill has the potential to increase academic achievement, improve self-care, reduce mortality and morbidity, and increase quality of life in this high risk, growing population.

ELIGIBILITY:
Inclusion Criteria:

* be 14-18 years old
* have SVHD
* undergone Fontan completion
* understands English
* able to read computer screen
* have phone access
* MoCA score of 25 to 10

Exclusion Criteria:

* pregnancy
* claustrophobia
* presence of loose metal
* prior head injury or stroke
* clinical diagnosis of depression
* previous cardiac arrest and ECMO use
* currently listed for heart transplant
* known genetic syndrome
* severe developmental delay
* born less than 35 weeks gestation

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in Working Memory Index [WMI] Scores | Baseline, 6 weeks
  To be measured by the Wide Range Assessment of Memory and Learning, version 2 [WRAML 2], working memory index [mean 100, SD 15] subscale. This is an administered test by trained personnel which measures all aspects of memory [visual, verbal, working memory, attention / concentration]. Lower scores indicate worse working memory deficits [1 SD below normal is < 85].

SECONDARY OUTCOMES:
Changes in Mean Diffusivity [MD] Values [brain tissue changes] | Baseline, 6 weeks
  To be measured non-invasively via brain MRI using diffusion tensor imaging (DTI) techniques, which measure mean diffusivity (MD) values (increased values indicate worse tissue injury).

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Pike, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA 300 Medical Plaza, Los Angeles, California, United States